CLINICAL TRIAL: NCT03083236
Title: A Randomised Controlled Trial of the Effectiveness of Parent-based Models of Speech and Language Therapy Intervention for 2 to 3 Year Old Children With Primary Language Delay in Areas of Social Disadvantage
Brief Title: Parent-based Intervention for Language Delayed 2 to 3 Year Olds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Solent NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Solent NHS Trust
Record Dates: First submitted 2017-03-08; First posted 2017-03-17 (Actual); Last update posted 2017-10-10 (Actual); Status verified 2017-10

CONDITIONS: Speech and Language Therapy
MeSH Terms: conditions — Communication Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Standard PBI — Standard Parent Based Intervention (PBI)
Other: Enhanced — Enhanced Parent Based Intervention (EPBI)

SUMMARY:
The aim of the study is to evaluate the impact of parent based intervention on the language of 2 to 3 year old children from socially disadvantaged populations with a clinical diagnosis of primary language delay.

DETAILED DESCRIPTION:
This project is original in proposing to evaluate the effectiveness of a parent-based intervention for a clinical population of 2 to 3 year olds with a diagnosis of primary language delay in areas of social disadvantage. It is original in developing an interagency, integrated model of delivery in line with the health and social care agenda (NHS 5 Year Forward Plan). It is also original in examining the effect of parent attitudes on child outcomes.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria (to diagnose primary language delay):

* The child is 24-36 months old
* The child has little or no expressive language (a vocabulary of 40 or less single words)
* The child has no known aetiology; the language delay is not secondary to sensory, structural, neurological or cognitive impairments
* The family have been assessed as having low socioeconomic status The study will use the Index of Multiple Deprivation (IMD) as a basis to determining a measure of deprivation. The IMD combines information from seven domains (income, employment, education, health, crime, housing and living environment) to produce an overall measure and it ranks how deprived areas are relative to others. This will be used to determine which areas and Children's Centres will be involved in the proposed RCT. However, as this is a geographical ranking, the RCT will include further refinement of eligibility of social disadvantage via assessment of individual measures of income deprivation, employment deprivation and education attainment. This information on employment and parent education levels will be collected via the case history taken at the initial assessment, as this is standard practice in a profile of risk for child language delay. The additional information on income will be taken at the first research assessment, as this does not form part of standard practice

Exclusion Criteria:

* The child's expressive language consists of a vocabulary of more than 40 single words
* The child's language delay is secondary to sensory, structural, neurological or cognitive impairments
* English is not the first language for the family.
* Where English is not the first language, children would be excluded. Adjustments to the protocol and delivery of intervention would be required where English is an additional language (EAL) and there is a need to test the intervention first on an English-speaking population. If effective, a longer term programme plan would be to amend the programme and evaluate the effectiveness with EAL children.

Ages: 24 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 192 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
The Pre-School Language Scales 5 UK (PLS 5 UK) | 2 years
  The planned primary outcome measure for the proposed RCT is a quantitative measure of child language using a standardised assessment measure, The Pre-School Language Scales 5 UK (PLS 5 UK) (Zimmerman et al, 2014). This will provide a sound measure of reliability and validity.

IPD SHARING:
Plan to Share IPD: No